CLINICAL TRIAL: NCT01745770
Title: Double-blind, Double-dummy, Randomised, Multi-centre, Comparative Phase III Clinical Study on the Efficacy and Tolerability of an 8 Week Oral Treatment With Three Times Daily 1000 mg Mesalazine Versus Three Times Daily 2x500 mg Mesalazine in Patients With Active Ulcerative Colitis
Brief Title: TID 1000 mg Mesalazine Versus TID 2x500 mg Mesalazine in Active Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAT-25/UCA
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Active Ulcerative Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Mesalazine - TID 1000 mg
- B (Active Comparator)
  Interventions: Drug: Mesalazine - TID 2x 500 mg

INTERVENTIONS:
Drug: Mesalazine - TID 1000 mg
  Arms: A
Drug: Mesalazine - TID 2x 500 mg
  Arms: B

SUMMARY:
The purpose of the trial is to proof whether TID 1000 mg mesalazine is non-inferior to TID 2x 500 mg mesalazine in the treatment of patients with acute ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men or women aged 18 to 75 years
* Active ulcerative colitis, except proctitis limited to 15 cm ab ano, confirmed by endoscopy and histology

Exclusion Criteria:

* Crohn's disease, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated colitis, microscopic colitis (i.e., collagenous colitis and lymphocytic colitis)
* Toxic megacolon
* Screening stool positive for germs causing bowel disease
* Malabsorption syndromes
* Celiac disease
* Other inflammatory or bleeding disorders of the colon and intestine, or diseases that may cause diarrhoea or gastrointestinal bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission | 8 weeks
  Proportion of patients with clinical remission at week 8 compared to baseline. Clinical remission includes normalisation of stool frequency and absence of blood in stools

SECONDARY OUTCOMES:
Number of stools per week | 8 weeks
Number of bloody stools per week | 8 weeks
Time to first resolution of clinical symptoms | 8 weeks
  Times to first resolution of symptoms defined as the periods from the day of first administration of trial medication , until the
  * First of at least 3 consecutive days each with =< 3 stools/day
  * First of at least 3 consecutive days each with no bloody stools/day,
  * First of at least 3 consecutive days each with =< 3 stools/day, all without blood

CONTACTS AND LOCATIONS:
Locations (1):
- Med. Klinik 1 - Markus-Krankenhaus, Frankfurt am Main, Hesse, Germany